CLINICAL TRIAL: NCT03300466
Title: A Randomized, Controlled, Evaluator-blinded, Split Face Study to Evaluate the Performance and Safety of GP0045 for Correction of Moderate to Severe Nasolabial Folds
Brief Title: A Study to Evaluate the Performance and Safety of GP0045 for Correction of Moderate to Severe Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43FE1630
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Results first posted 2020-04-17 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2020-04

CONDITIONS: Nasolabial Fold; Safety
Keywords: Hyaluronic Acid, Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP0045 (Experimental): Treatment with GP0045
  Interventions: Device: GP0045
- Comparator (Active Comparator): Treatment with active comparator
  Interventions: Device: Comparator

INTERVENTIONS:
Device: GP0045 — Hyaluronic acid gel
  Arms: GP0045
Device: Comparator — Hyaluronic acid gel
  Arms: Comparator

SUMMARY:
This is a study to assess the performance and safety of GP0045 when injected in the nasolabial folds.

There is an 18 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Ability to adequately understand the verbal explanations and the written subject information provided in local language and ability to give consent to participate in the study
* Signed and dated informed consent to participate in the study, including photo consent
* Subjects with intent to undergo correction of both nasolabial folds

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel
* Known/previous allergy or hypersensitivity to local anesthetics, e.g. lidocaine or other amide-type anesthetics
* Any condition (medical or other) that, in the opinion of the Investigator, would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may interfere with the outcome of the study)
* Participation in any other clinical study with an investigational product within 30 days before treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (1):
- Q-Med, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- GP0045 in Right NLF and Comparator in Left NLF: Treatment with GP0045 in right NLF (nasolabial fold) and comparator in left NLF
  GP0045: Hyaluronic acid gel Comparator: Hyaluronic acid gel
- Comparator in Right NLF and GP0045 in Left NLF: Treatment with comparator in right NLF and GP0045 in left NLF
  GP0045: Hyaluronic acid gel Comparator: Hyaluronic acid gel
Period: Overall Study
Arm/Group | GP0045 in Right NLF and Comparator in Left NLF | Comparator in Right NLF and GP0045 in Left NLF
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GP0045 in Right NLF and Comparator in Left NLF: Treatment with GP0045 in right NLF and comparator in left NLF
  GP0045: Hyaluronic acid gel Comparator: Hyaluronic acid gel
- Total: Total of all reporting groups
Arm/Group | GP0045 in Right NLF and Comparator in Left NLF | Comparator in Right NLF and GP0045 in Left NLF | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Response Rate in Treatment of Nasolabial Fold (NLF) Based on a Scale
Description: The scale is a 5-graded NLF wrinkle severity scale ranging from absent (Grade 1) to severe (Grade 5). The response rate was defined as the percentage of subjects with at least 1 grade improvement in NLF wrinkle severity. Assessment made by blinded evaluator.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Groups:
- Comparator: Treatment with comparator
  Comparator: Hyaluronic acid gel
Arm/Group | GP0045 | Comparator
Number analyzed (Participants) | 19 | 19
percentage of participants | 63.2 | 68.4

2. Secondary Outcome: Response Rate in Treatment of Nasolabial Fold (NLF) Based on a Scale
Description: as for outcome 1
Time Frame: 2 weeks, 3, 9, 12, 15 and 18 months
Measure: Number; unit: percentage of participants
Arm/Group | GP0045 | Comparator
Number analyzed (Participants) | 19 | 19
percentage of participants
  2 weeks | 100 | 100
  3 months | 89.5 | 89.5
  9 months | 36.8 | 26.3
  12 months | 15.8 | 21.1
  15 months | 10.5 | 5.3
  18 months | 0 | 0

ADVERSE EVENTS:
Time Frame: 18-19 months (depending on how long screening), from screening visit to final study visit.
Groups:
- GP0045 in Right NLF and Comparator in Left NLF: Treatment with GP0045 in right NLF (nasolabial fold) and comparator in left NLF
- Comparator in Right NLF and GP0045 in Left NLF: Treatment with comparator in right NLF and GP0045 in left NLF
Arm/Group | GP0045 in Right NLF and Comparator in Left NLF | Comparator in Right NLF and GP0045 in Left NLF
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP0045 in Right NLF and Comparator in Left NLF (N=10) | Comparator in Right NLF and GP0045 in Left NLF (N=10)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to study product/study product injection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP0045 in Right NLF and Comparator in Left NLF (N=10) | Comparator in Right NLF and GP0045 in Left NLF (N=10)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (2) — Related to study product or injection procedure. One event in right NLF (treated with comparator) and one event in left NLF (treated with GP0045).
Implant site erythema (General disorders) | 0 (0) | 1 (2) — Related to study product or injection procedure. One event in right NLF (treated with comparator) and one event in left NLF (treated with GP0045).
Implant site hypoesthesia (General disorders) | 0 (0) | 1 (1) — Related to study product or injection procedure. In left NLF (treated with GP0045).
Implant site mass (General disorders) | 1 (1) | 1 (1) — Related to study product or injection procedure. Both events in the NLF treated with GP0045.
Implant site pain (General disorders) | 0 (0) | 7 (17) — Related to study product/injection. 9 events (5 participants) in the NLF treated with GP0045, 8 events (4 participants) in the NLF treated with comparator. (1 participant can report one event in left NLF and one event in right NLF at the same time.)
Implant site papules (General disorders) | 0 (0) | 1 (1) — Related to study product or injection procedure. In the NLF treated with GP0045.
Implant site pruritus (General disorders) | 0 (0) | 1 (2) — Related to study product or injection procedure. One event in the NLF treated with GP0045 and one event in the NLF treated with comparator.
Implant site swelling (General disorders) | 0 (0) | 4 (11) — Related to study product/injection. 9 events (3 participants) in NLF treated with GP0045, 2 events (2 participants) in the NLF treated with comparator. (1 participant can report 1 event in the right NLF and 1 event in the left NLF at the same time).
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Eye allergy (Eye disorders) | 1 (1) | 0 (0) — Unrelated to study product/study product injection
Iritis (Eye disorders) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated to study product/study product injection
Gingival recession (Gastrointestinal disorders) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Toothache (Gastrointestinal disorders) | 3 (3) | 0 (0) — Unrelated to study product/study product injection
Nodule (General disorders) | 0 (0) | 1 (2) — Unrelated to study product/study product injection
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) — Unrelated to study product/study product injection
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Influenza (Infections and infestations) | 2 (2) | 0 (0) — Unrelated to study product/study product injection
Nasopharyngitis (Infections and infestations) | 5 (5) | 7 (8) — Unrelated to study product/study product injection
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) — Unrelated to study product/study product injection
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Unrelated to study product/study product injection
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) — Unrelated to study product/study product injection
Urinary tract infection (Infections and infestations) | 1 (4) | 0 (0) — Unrelated to study product/study product injection
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Unrelated to study product/study product injection
Overweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Unrelated to study product/study product injection
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Unrelated to study product/study product injection
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated to study product/study product injection
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to study product/study product injection
Headache (Nervous system disorders) | 3 (5) | 4 (9) — Unrelated to study product/study product injection
Hematoma (Vascular disorders) | 1 (1) | 0 (0) — Unrelated to study product/study product injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT03300466/Prot_SAP_000.pdf